CLINICAL TRIAL: NCT05292313
Title: Pilot for Dual Implant Versus Single Implant Distal End of Femur (pDISIDE Femur)
Brief Title: Dual Implant Versus Single Implant Distal End of Femur
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Justin Haller, Principle Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 149119
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Distal Femur Fracture
Keywords: Distal Femur Fracture; Dual distal femur implants; Single distal femur implant; Mortality
MeSH Terms: conditions — Femoral Fractures, Distal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single distal femur implant (Other): Single implant constructs will be either a retrograde intramedullary nail with interlocking screws or a single plate and screw construct.
  Interventions: Procedure: Single distal femur implant
- Dual distal femur implants (Other): Dual implant constructs will either be an intramedullary nail with an additional plate and screw construct or dual (two plates in any orientation) plate and screw construct.
  Interventions: Procedure: Dual distal femur implants

INTERVENTIONS:
Procedure: Single distal femur implant — Single implant fixation
  Arms: Single distal femur implant
Procedure: Dual distal femur implants — Dual implant fixation
  Arms: Dual distal femur implants

SUMMARY:
The investigators overall study objective is to determine the difference in outcomes for patients over 60 years of age with a displaced distal femur fracture treated with dual distal femur implants (dual plate or IMN/plate) vs. a single distal femur implant (plate or IMN).

DETAILED DESCRIPTION:
The incidence of distal femur fractures in elderly patients continues to increase, most recently having an incidence of 8.7/100,000/year. This trend likely accompanies the aging population and the increased rates of knee arthroplasty. While these fractures are far less common than geriatric hip fractures, distal femur fractures present similar treatment challenges. Elderly distal femur fractures tend to occur in compromised hosts with poor bone mineral density. Similar to geriatric hip fractures, care emphasizes early mobilization to avoid the complications associated recumbency, including pneumonia, pressure sores, and venous thromboembolism. These patients are often unable to mobilize with restricted weight bearing, which places significant stress on the fixation construct. As a result, elderly patients with distal femur fractures can have high rates of morbidity and mortality.

Despite several prior studies reporting one year mortality greater than 20%, elderly distal femur fractures do not receive the same attention as geriatric hip fractures. These patient injuries are likely similar in terms of their age and comorbidities while having the same issues with post-operative mobility. Therefore, it makes sense that geriatric distal femur fracture patients and geriatric hip fracture patients have similar mortality rates. Investigators recently reported significantly greater in-hospital mortality in geriatric distal femur fractures as compared to geriatric hip fractures. A recent study of the US Medicare database is the largest study on geriatric distal femur fractures in the literature, and the overall mortality of 18.5% is similar to several prior studies ranging from 13-38%.

Distal femur fractures have traditionally been treated with operative fixation using either a lateral plate or an intramedullary nail. Advances in plate and nail technology allow for distal femur fractures to be stabilized with minimal soft tissue dissection. While recent studies suggest that early weight bearing can be tolerated with low failure rates, many surgeons continue to institute weight-bearing restrictions for osteopenic patients treated with operative fixation. Nonunion rates for operatively treated distal femur fractures have been reported to be as high as 20% in large series, leading to additional surgery to achieve union. These limitations with operative fixation have led surgeons to investigate the utility of supplementing the fixation with additional plates and/or nails.

Since many surgeons may not allow early weight bearing in osteopenic patients with operatively treated distal femur fractures, dual plating of the distal femur and locked plate/IMN combinations have become increasingly popular. Biomechanical studies have demonstrated increased torsional stiffness and axial stiffness in dual plate and plate/nail constructs as compared to single implant. A recent meta-analysis by other investigators has further demonstrated dual implants for distal femur fractures to have a low complication rate (5% nonunion) as compared to prior evidence of single implant fixation (0-25% nonunion).

In the recent study, authors reported a trend toward less one year mortality in patients treated with distal femoral replacement (DFR) (13.8%) as compared to operative fixation (22.6%) despite finding similar mortality rates at 90 days post-operatively. Since the complication rate was significantly greater in the DFR cohort, this one year mortality benefit is presumably related to early patient weight bearing after DFR that may not be permitted as frequently with operative fixation. Additionally, patients with a DFR may achieve more early mobility than operatively treated patients who are permitted immediate weight bearing due to enhanced stability in the DFR construct. Using dual implants to treat distal femur fractures may allow patients to achieve early mobility and similar mortality as a DFR patients, but have fewer post-surgical complications and less cost than a DFR.

The investigators overall study aim is to determine the difference in outcomes for patients over 60 years of age with a displaced distal femur fracture treated with dual distal femur implants (dual plate or IMN/plate) vs. a single distal femur implant (plate or IMN).

ELIGIBILITY:
Inclusion Criteria:

* Patient age 60 years or greater,
* Femur fracture distal to the femoral diaphysis,
* Operative treatment within 72 hours of presenting to the treating hospital,
* Patient was previously ambulatory,
* Fracture amendable to either single or dual implant fixation,
* Informed consent can be obtained from the patient, family member, or power of attorney.

Exclusion Criteria:

* Associated major lower extremity fracture,
* Ongoing infection,
* History of metabolic bone disease (Paget's, etc),
* Pathologic fracture,
* Open fracture,
* Severe cognitive impairment (Six Item Screener with 3 or more errors),
* Stage 5 Parkinson's disease,
* Significant femoral bone loss requiring planned staged bone grafting,
* Vascular injury.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1-year
  The primary outcome will be one-year mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Haller, M.D., Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No